CLINICAL TRIAL: NCT02063867
Title: Cluster-Randomized Controlled Trial of Hospitals to Reduce Healthcare-Associated Infections and Readmissions Through Routine Bathing With Antiseptic Soap and Targeted Use of Nasal Antibiotic Ointment (ABATE Infection Trial)
Brief Title: Active Bathing to Eliminate Infection (ABATE Infection) Trial
Acronym: ABATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Harvard Pilgrim Health Care (Other); Hospital Corporation of America (Industry); Rush University (Other); Cook County Health (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Susan Huang, Associate Professor and Medical Director of Epidemiology and Infection Prevention, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 367981; UH2AT007769 (NIH); UH3AI113337 (NIH)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-06

CONDITIONS: Healthcare Associated Infections; Methicillin Resistant Staphylococcus Aureus; Multi Drug Resistant Organisms
Keywords: HAI; MRSA; VRE
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Usual Care (No Intervention): Routine policy for showering or bathing non-critical care patients
- Arm 2: Decolonization (Active Comparator): Daily chlorhexidine (CHG) shower or CHG cloth bath for all non-critical care patients.
  Topical intranasal mupirocin ointment (bilateral nares, twice daily) x5 days if non-critical care patients are MRSA+ by history, culture, or screen.
  Interventions: Drug: Arm 2: Decolonization

INTERVENTIONS:
Drug: Arm 2: Decolonization — Daily chlorhexidine (CHG) shower or CHG cloth bath for all non-critical care patients.
  Topical intranasal mupirocin ointment (bilateral nares, twice daily) x5 days if non-critical care patients are MRSA+ by history, culture, or screen.
  Arms: Arm 2: Decolonization

SUMMARY:
The ABATE Infection Project is a cluster randomized trial of hospitals to compare two quality improvement strategies to reduce multi-drug resistant organisms and healthcare-associated infections in non-critical care units. The two strategies to be evaluated are:

* Arm 1: Routine Care Routine policy for showering/bathing
* Arm 2: Decolonization Use of chlorhexidine as routine soap for showering or bed bathing for all patients Mupirocin x 5 days if MRSA+ by history, culture, or screen

Note that enrolled "subjects" represents 53 individual HCA Hospitals (representing ~190 non-critical care units) that have been randomized.

ELIGIBILITY:
Inclusion Criteria:

* All HCA hospitals that reside in the United States
* Note: Unit of randomization is the hospital, but the participants are hospital units

Exclusion Criteria:

* Non-critical care units where chlorhexidine bathing or decolonization for MRSA+ non-critical care patients is routine
* Pediatric, peri-partum, rehabilitation, psychiatry, and BMT units
* Units with >30% cardiac or hip/knee orthopedic surgeries
* Unit average length of stay <2 days
* Patients <12 years-old
* Patients with known allergy to mupirocin or chlorhexidine

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-04; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Huang, MD MPH, Principal Investigator — University of California, Irvine; Ken Kleinman, ScD, Study Director — University of Massachusetts, Amherst; Edward Septimus, MD, Study Director — Hospital Corporation of America; Jason Hickok, MBA, RN, Study Director — Hospital Corporation of America; Julia Moody, MS, Study Director — Hospital Corporation of America; Mary Hayden, MD, Study Director — Rush University; Robert Weinstein, MD, Study Director — John Stroger Hospital; John Jernigan, MD MS, Study Director — Centers for Disease Control and Prevention; Jonathan Perlin, MD PhD, Study Director — Hospital Corporation of America; Daniel Gillen, PhD, Study Director — University of California, Irvine; Grace Lee, MD MPH, Study Director — Harvard Pilgrim Health Care Institute
Locations (52):
- United States (52):
  - West Hills Hospital & Medical Center, West Hills, California
  - North Suburban Medical Center, Thornton, Colorado
  - Blake Medical Center, Bradenton, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Palms West Hospital, Loxahatchee Groves, Florida
  - Orange Park Medical Center, Orange Park, Florida
  - West Florida Hospital, Pensacola, Florida
  - Northside Hospital, St. Petersburg, Florida
  - St. Petersburg General Hospital, St. Petersburg, Florida
  - South Bay Hospital, Sun City Center, Florida
  - West Palm Hospital, West Palm Beach, Florida
  - Cartersville Medical Center, Cartersville, Georgia
  - Coliseum Northside Hospital, Macon, Georgia
  - Eastside Medical Center, Snellville, Georgia
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Regional Medical Center of Acadiana, Lafayette, Louisiana
  - Garden Park Medical Center, Gulfport, Mississippi
  - Research Medical Center, Kansas City, Missouri
  - Lee's Summit Medical Center, Lee's Summit, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - MountainView Hospital-Las Vegas, Las Vegas, Nevada
  - Parkland Medical Center, Derry, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Colleton Medical Center, Walterboro, South Carolina
  - Parkridge Medical Center, Chattanooga, Tennessee
  - Parkridge East Hospital, Chattanooga, Tennessee
  - TriStar Horizon Medical Center, Dickson, Tennessee
  - Hendersonville Medical Center, Hendersonville, Tennessee
  - Summit Medical Center, Hermitage, Tennessee
  - St. David's Medical Center, Austin, Texas
  - Valley Regional Medical Center, Brownsville, Texas
  - Conroe Regional Medical Center, Conroe, Texas
  - Corpus Christi Medical Center, Corpus Christi, Texas
  - Las Palmas Medical Center, El Paso, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - Las Colinas Medical Center, Irving, Texas
  - Kingwood Medical Center, Kingwood, Texas
  - Northeast Methodist Hospital, Live Oak, Texas
  - Rio Grande Regional Hospital, McAllen, Texas
  - North Hills Hospital, North Richland Hills, Texas
  - Medical Center of Plano, Plano, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - Methodist Stone Oak Hospital, San Antonio, Texas
  - Clear Lake Regional Medical Center, Webster, Texas
  - Timpanogos Regional Hospital, Orem, Utah
  - John Randolph Medical Center, Hopewell, Virginia
  - LewisGale Hospital-Alleghany, Low Moor, Virginia
  - Reston Hospital Center, Reston, Virginia
  - Chippenham Johnston Willis Medical Center, Richmond, Virginia
  - Henrico Doctors' Hospital, Richmond, Virginia

REFERENCES:
- [Derived] Huang SS, Septimus E, Kleinman K, Moody J, Hickok J, Heim L, Gombosev A, Avery TR, Haffenreffer K, Shimelman L, Hayden MK, Weinstein RA, Spencer-Smith C, Kaganov RE, Murphy MV, Forehand T, Lankiewicz J, Coady MH, Portillo L, Sarup-Patel J, Jernigan JA, Perlin JB, Platt R; ABATE Infection trial team. Chlorhexidine versus routine bathing to prevent multidrug-resistant organisms and all-cause bloodstream infections in general medical and surgical units (ABATE Infection trial): a cluster-randomised trial. Lancet. 2019 Mar 23;393(10177):1205-1215. doi: 10.1016/S0140-6736(18)32593-5. Epub 2019 Mar 5. PMID 30850112
- [Derived] Johnson KE, Neta G, Dember LM, Coronado GD, Suls J, Chambers DA, Rundell S, Smith DH, Liu B, Taplin S, Stoney CM, Farrell MM, Glasgow RE. Use of PRECIS ratings in the National Institutes of Health (NIH) Health Care Systems Research Collaboratory. Trials. 2016 Jan 16;17:32. doi: 10.1186/s13063-016-1158-y. PMID 26772801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Participant Flow section reflects numbers of hospitals that were enrolled in the intervention (the unit of enrollment and randomization was hospital), as well as the number of participants included in analysis, (the number of patient admissions from participating units in the enrolled hospitals), in each arm during the intervention period.
Units Other Than Participants: hospitals
Groups:
- Arm 2: Decolonization: Daily chlorhexidine (CHG) shower or CHG cloth bath for all non-critical care patients.
  Topical intranasal mupirocin ointment (bilateral nares, twice daily) x5 days if non-critical care patients are MRSA+ by history, culture, or screen.
  Arm 2: Decolonization: Daily chlorhexidine (CHG) shower or CHG cloth bath for all non-critical care patients.
  Topical intranasal mupirocin ointment (bilateral nares, twice daily) x5 days if non-critical care patients are MRSA+ by history, culture, or screen.
Period: Overall Study
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Started | 156889; 26 hospitals | 183013; 27 hospitals
Completed | 152598; 24 hospitals | 180048; 24 hospitals
Not Completed | 4291; 2 hospitals | 2965; 3 hospitals

BASELINE CHARACTERISTICS:
Population: These numbers reflect the number of participants in the baseline period across all participating facilities enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization | Total
Number analyzed (Participants) | 156889 | 183013 | 339902
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (18.2) | 62.6 (18.6) | 62.4 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not available for 32 patients during the intervention period.
  Participants
    number analyzed (Participants) | 156873 | 182997 | 339870
    Female | 84585 | 100249 | 184834
    Male | 72288 | 82748 | 155036
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 107261 | 112067 | 219328
  Hispanic | 22581 | 38704 | 61285
  Black | 21501 | 22462 | 43963
  Asian | 2021 | 4175 | 6196
  Other/Unknown | 3525 | 5605 | 9130
Region of Enrollment [Number; unit: participants]
  United States | 156889 | 183013 | 339902

OUTCOME MEASURES:

1. Primary Outcome: MRSA and VRE Clinical Cultures
Description: Methicillin-resistant Staphylococcus aureus (MRSA) and vancomycin-resistant enterococci (VRE) clinical cultures attributable to participating units. Defined as occurring >2 days into a participating unit stay through 2 days following unit discharge
Time Frame: 21 months
Population: Unadjusted intention-to-treat analysis. Number of patients in the intervention period provided. Analysis involves comparison of baseline and intervention patients (difference in differences)
Measure: Number (95% Confidence Interval); unit: Hazard Ratio (Intervention vs Baseline)
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Number analyzed (Participants) | 156889 | 183013
Hazard Ratio (Intervention vs Baseline) | 0.87 [0.79 to 0.95] | 0.79 [0.73 to 0.87]
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Decolonization; Test type: Superiority; p = 0.17, Mixed Models Analysis; Assessed if hazard ratio between intervention vs baseline periods differs between study groups, accounting for clustering within hospitals

2. Secondary Outcome: Gram-negative Multi-drug Resistant Organism Clinical Cultures
Description: Gram-negative (GN) multi-drug resistant organism clinical cultures attributable to participating units. Defined as occurring >2 days into a participating unit stay through 2 days following unit discharge
Time Frame: 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio (Intervention vs Baseline)
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Number analyzed (Participants) | 156889 | 183013
Hazard Ratio (Intervention vs Baseline) | 0.81 [0.72 to 0.91] | 0.91 [0.82 to 1.00]
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Decolonization; Test type: Superiority; p = 0.16, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: All-cause Bloodstream Infections
Description: All-cause bloodstream infections attributable to participating units. Defined as occurring >2 days into a participating unit stay through 2 days following unit discharge. Includes bacterial and yeast pathogens. Skin commensals require two positive blood cultures.
Time Frame: 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Number analyzed (Participants) | 156889 | 183013
Hazard Ratio | 0.96 [0.85 to 1.08] | 0.90 [0.80 to 1.01]
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Decolonization; Test type: Superiority; p = 0.43, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Urinary Tract Infections
Description: Urinary tract infections attributable to participating units. Defined as occurring >2 days into a participating unit stay through 2 days following unit discharge
Time Frame: 21 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Blood Culture Contamination
Description: Blood culture contamination
Time Frame: 21 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Clostridium Difficile Infection
Description: Clostridium difficile Infection attributable to participating units
Time Frame: 21 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: 30-Day Infectious Readmissions
Description: 30-Day Infectious Readmissions among patients in participating units
Time Frame: 21 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Emergence of Resistance to Chlorhexidine or Mupirocin
Description: Emergence of resistance to chlorhexidine (among MRSA and select gram-negative bacteria) or mupirocin (among MRSA) for strains isolated from participating units
Time Frame: 21 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Cost Effectiveness
Description: Cost effectiveness of routine care vs decolonization
Time Frame: 21 months
Reporting Status: Not Posted

10. Post Hoc Outcome: MRSA and VRE Clinical Cultures Among Patients With Devices
Description: Sub-population analysis: Methicillin-resistant Staphylococcus aureus (MRSA) and vancomycin-resistant enterococci (VRE) clinical cultures attributable to participating units (defined as occurring >2 days into a participating unit stay through 2 days following unit discharge), among patients with medical devices (central venous catheters (including accessed ports), midline catheters, or lumbar drains).
Time Frame: 21 months
Population: Unadjusted intention-to-treat analysis of sub-population: patients with medical devices (central venous catheters (including accessed ports), midline catheters, or lumbar drains). Number of patients in the intervention period provided. Analysis involves comparison of baseline and intervention patients (difference in differences)
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Number analyzed (Participants) | 15372 | 23417
Hazard Ratio | 1.17 [1.00 to 1.37] | 0.80 [0.69 to 0.92]
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Decolonization; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

11. Post Hoc Outcome: MRSA Clinical Cultures Among Patients With Devices
Description: Sub-population analysis: Methicillin-resistant Staphylococcus aureus (MRSA) clinical cultures attributable to participating units (defined as occurring >2 days into a participating unit stay through 2 days following unit discharge), among patients with medical devices (central venous catheters (including accessed ports), midline catheters, or lumbar drains).
Time Frame: 21 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Number analyzed (Participants) | 15372 | 23417
Hazard Ratio | 1.17 [0.99 to 1.39] | 0.87 [0.74 to 1.02]
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Decolonization; Test type: Superiority; p = 0.0126, Mixed Models Analysis — Remains significant after adjusting for multiple comparisons; [statistical method as in outcome 1, analysis 1]

12. Post Hoc Outcome: VRE Clinical Cultures Among Patients With Devices
Description: Sub-population analysis: Vancomycin-resistant enterococci (VRE) clinical cultures attributable to participating units (defined as occurring >2 days into a participating unit stay through 2 days following unit discharge), among patients with medical devices (central venous catheters (including accessed ports), midline catheters, or lumbar drains).
Time Frame: 21 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Number analyzed (Participants) | 15372 | 23417
Hazard Ratio | 1.26 [0.85 to 1.86] | 0.58 [0.44 to 0.78]
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Decolonization; Test type: Superiority; p = 0.002, Mixed Models Analysis — Remained significant after adjusting for multiple comparisons; [statistical method as in outcome 1, analysis 1]

13. Post Hoc Outcome: All-cause Bloodstream Infections Among Patients With Devices
Description: Sub-population analysis: All-cause bloodstream infections attributable to participating units (defined as occurring >2 days into a participating unit stay through 2 days following unit discharge), among patients with medical devices (central venous catheters (including accessed ports), midline catheters, or lumbar drains). Includes bacterial and yeast pathogens. Skin commensals require two positive blood cultures.
Time Frame: 21 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
Number analyzed (Participants) | 15372 | 23417
Hazard Ratio | 1.13 [0.96 to 1.33] | 0.81 [0.70 to 0.94]
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Decolonization; Test type: Superiority; p = 0.0032, Mixed Models Analysis — Remained significant after adjusting for multiple comparisons; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Intervention duration (21 months)
Arm/Group | Arm 1: Usual Care | Arm 2: Decolonization
All-Cause Mortality (participants affected / at risk) | 0/156889 | 0/183013
Serious Adverse Events (participants affected / at risk) | 0/156889 | 0/183013
Other Adverse Events (participants affected / at risk) | 0/156889 | 25/183013
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Usual Care (N=156889) | Arm 2: Decolonization (N=183013)
Diffuse rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Diffuse itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild rash on trunk (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Mild rash, location unknown (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild rash on limbs (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Mild rash on limbs, trunk (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Mild rash on groin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild rash on limbs, face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild rash on limbs, groin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild rash on limbs, trunk, face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild rash on limbs, trunk, groin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild rash on neck, forehead (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT02063867/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT02063867/SAP_001.pdf